CLINICAL TRIAL: NCT04238845
Title: Assessment of a Combined Strategy of Seasonal Malaria Chemoprevention + Supplementation With PlumpyDoz and Vitamin A-Zinc to Prevent Malaria and Malnutrition in Burkina Faso
Brief Title: Assessment of a Combined Strategy of SMC + Nutrients Supplementation to Tackle Malaria and Malnutrition
Acronym: SMC-NUT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TMA2018CDF-2365
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-03

CONDITIONS: Malaria; Malnutrition, Child
Keywords: Malaria; Malnutrition; Chemoprevention
MeSH Terms: conditions — Malaria; Child Nutrition Disorders; Malnutrition | interventions — Dietary Supplements; Vitamin A; Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SMC + Vitamin A alone (Active Comparator): Children under SMC Coverage, receiving AQSP and Vitamin A supplementation alone
  Interventions: Drug: AQSP Administration; Dietary Supplement: Supplementation with Vitamin A
- SMC+ Vitamin A + Plumpy'Doz (Experimental): Children under SMC Coverage, receiving AQSP + Vitamin A plus Plumpy'Doz supplementation
  Interventions: Drug: AQSP Administration; Dietary Supplement: Supplementation with Plumpy'Doz; Dietary Supplement: Supplementation with Vitamin A
- SMC+ Vitamin A + Zinc (Experimental): Children under SMC Coverage, receiving AQSP + Vitamin A plus Zinc supplementation
  Interventions: Drug: AQSP Administration; Dietary Supplement: Supplementation with Vitamin A; Dietary Supplement: Supplementation with Zinc

INTERVENTIONS:
Drug: AQSP Administration — Three days treatment of all children with AQSP for SMC
Dietary Supplement: Supplementation with Plumpy'Doz — Daily supplementation of children with Plumpy'Doz
  Arms: SMC+ Vitamin A + Plumpy'Doz
Dietary Supplement: Supplementation with Vitamin A — Single dose supplementation with Vitamin A to all children
Dietary Supplement: Supplementation with Zinc — Daily supplementation with Zinc
  Arms: SMC+ Vitamin A + Zinc

SUMMARY:
Malaria and malnutrition represent major public health concerns worldwide especially in Sub-Sahara Africa. Despite implementation of Seasonal Malaria Chemoprophylaxis (SMC), an intervention aimed at reducing malaria prevalence among children aged 6- 59 months, the burden of malaria and associated mortality among children below age 5 years remains high in Burkina Faso. This raises the question of what hiding factors may negatively affect the responsiveness of SMC intervention. Malnutrition, in particular micronutrient deficiency, is one of these potential factors that can negatively affect the effectiveness of SMC. Treating micronutrient deficiencies is known to reduce the prevalence of malaria mortality in highly prevalent malaria zone such as rural settings. Therefore, the hypothesis that a combined strategy of SMC together with a daily oral nutrients supplement (Vitamin A-Zinc OR fortified peanut butter-like paste-Plumpy'Doz) will enhance the immune response and decrease the incidence of malaria in this population and at the same time reduce the burden of malnutrition among children under SMC coverage was postulated.

Prior to the SMC implementation by the National Malaria Control Program (NMCP), children under SMC coverage will be identified through the Health and Demographic Surveillance System (HDSS). Children will be randomly assigned to one of the three groups (a) SMC + Vitamin A alone, (b) SMC + Vitamin A+ Zinc, or (c) SMC+Vitamin A + Plumpy'Doz. After each SMC monthly distribution, children will be visited at home to confirm drug administration and follow-up for one year. Anthropometric indicators will be recorded at each visit. Blood samples will be collected for thick and thin film and hemoglobin measurement and spotted onto filter paper for further PCR analyses.

This project will serve as a pilot of an integrated strategy in order to mutualize resources for best impact. By relying on existing strategies, the policy implementation of this joint intervention will be scalable at country and regional levels.

DETAILED DESCRIPTION:
Malaria is hyper-endemic in Burkina Faso and many sub-Saharan Africa countries. According to the National Malaria Control Program (NMCP) approximately 11 915 816 malaria cases and 4 144 malaria-related deaths were reported in 2017 in Burkina Faso. Numerous malaria control interventions have been implemented in Burkina Faso in order to achieve the 2030 Sustainable Development Goal (SDG) 3. Seasonal malaria chemo-prevention (SMC) ranks among the largest and reliable interventions for malaria control in countries with marked seasonality of malaria transmission. This preventive measures involves administering antimalarial drugs (Amodiaquine-Sulfadoxine-Pyrimethamine) to children aged 6- 59 months on a monthly basis during the high transmission peak. In Burkina Faso, SMC is implemented from July/August to October/November each year. SMC is recommended by the World Health Organization (WHO) and is known to reduce malaria morbidity by 30 to 80%. Despite the implementation of this strategy, the burden of malaria and associated mortality is still very high in this population in Burkina Faso. This raises questions about other hidden factors that can negatively affect the effectiveness of SMC intervention.

At the same time, malnutrition is a major cause of childhood morbidity and mortality in low- and middle-income countries such as Burkina Faso. Malnutrition can lower immune system leading to increased severity of malaria in the population. The National Nutrition Program (NPP), which is the agency established to address malnutrition problems in Burkina Faso, currently aims to scale-up Community Management of Acute Malnutrition (CMAM). Both malaria and malnutrition are highly prevalent in rural settings. Furthermore, malaria seasonal peak coincides with period of food crisis in the country suggesting that malnutrition may influence malaria incidence during that period. Children under five years again represent the most vulnerable group. Importantly, treating micronutrient deficiencies is known to reduce malaria morbidity and mortality. Plumpy'Doz is specifically formulated for prevention of malnutrition in children from 6 months of age and adults. It has been recommended since 2007 by the WHO, UN Children's Fund (UNICEF), World Food Program (WFP), and the UN Standing Committee on Nutrition in the joint declaration on community-based management of severe acute malnutrition. Evidence also shows that Vitamin A-Zinc supplementation reduce malaria morbidity. A reduction by 20-30% of malaria incidence through micronutrient supplementation such as Vitamin A-Zinc has also been reported.

These aspects underlie the idea of the SMC-Nutrition project. This combined strategy could enhance the immune response and therefore decrease the severity of malaria in this population and at the same time reduce the burden of malnutrition in children under SMC coverage. This project will serve as a pilot integrated strategy in order to mutualize resources for best impact. By relying on existing strategies, the policy implementation of this joint intervention will be scalable at country and regional levels. If the pilot produces promising results, a large-scale multi-centric assessment of the strategy will be performed in several SMC countries (i.e. Niger, Mali and Burkina Faso).

Purpose and objective(s) Aim 1: To assess the feasibility of combining two different strategies led by different programs (malaria and nutrition) which affect the same target population (children under five years). SMC is a larger community-based intervention at a national level led by the NMCP. National Nutrition Program is trying to scale up the Community Management of Acute Malnutrition (CMAM). This project will serve as a pilot of integrated strategy in order to mutualize resources for best impact. By relying on existing strategies, the policy implementation of this joint intervention will be scalable at country and regional levels.

Aim 2: To boost the impact of SMC intervention in terms of reducing malaria morbidity, mortality and reduce the burden of malnutrition and anaemia in children under five years through supplementation with micronutrients and Vitamin A-Zinc.

Primary objectives 1: to assess in a randomized superiority trial whether SMC + Vitamin A+ Zinc or SMC+ Vitamin A+ Plumpy'Doz is more effective and safe in reducing uncomplicated malaria incidence, severe malaria incidence and related mortality compared to the SMC+ Vitamin A alone Primary objectives 2: to investigate the impact of the combined strategy in reducing the burden of malnutrition through reduction of anaemia incidence, mid-upper arm circumference gain, and weight gain.

Secondary objectives 1: to assess the impact of each treatment arm on the circulation parasite population through monitoring the temporal trend of antimalarial resistance molecular markers pfcrt, pfmdr1, dhfr and dhps.

Secondary objectives 2: to assess the coverage and compliance to SMC in the study area.

Secondary objectives 3: to determine the overall risk of adverse events (AEs).

Study population The target population is children under five years under SMC coverage and living across HDSS area

Subgroup analysis Three subgroups will be defined: (i) SMC + Vitamin A alone (ii) SMC+ Vitamin A+ Zinc and (iii) SMC+ Vitamin A +Plumpy'Doz

Proposed sample size The overall sample size for the study was estimated at 882 (3×294) to detect a 10% difference in risk of malaria occurrence between SMC alone group and any of SMC+ supplement group. Further assuming that 20% of the individuals will be lost to follow-up, an adjusted sample size of 353 children per arm was required. The final estimated sample size for this study is thus 1,059 children.

Trial design This is post-marketing phase. All the products that will be used in this study are recommended by WHO and are already used as part of routine management of acute malnutrition in Burkina Faso. Eligible children will be assigned to one of the three study arms: (i) SMC + Vitamin A alone (ii) SMC+ Vitamin A + Zinc and (iii) SMC+ Vitamin A + Plumpy'Doz. Administration of Amodiaquine-Sulfadoxine Pyrimethamine (AQ-SP) will not be performed by the study team but by the NMCP.

Randomisation method A computer-based randomization system will be used to assign the included children. The allocation will be performed at a central level (pharmacie of the CRUN) by the pharmacist phone call (pharmacist-field workers) following the inclusion number.

Protection against sources of bias This will be an open label study. No blinding is planned. However, to avoid contamination, only one child per household will be included.

Study duration Enrolment of participants will be implemented in parallel with SMC implementation by the National Malaria Control Program (NMCP). The randomized children will be followed-up actively for 6 Months and passively for six months to fully cover the high and low transmission periods.

Product(s) to be tested All the products that will be used in this study are recommended by WHO and are already used as part of routine management of acute malnutrition in Burkina Faso. The study products include Vitamin A-Zinc and Plumpy'Doz. Administration of Amodiaquine-Sulfadoxine Pyrimethamine (AQSP) will not be performed by the study team. SMC is implemented by the NMCP and all children 6-59 months are expected to be covered. Vitamin A supplemention will be performed by the Direction of Nutrition as a nationalwide campaign for the prevention of malnutrition in children under five years of age.

Product supply The product will be supplied to the household fortnightly. The stock will be ordered from accredited manufacturer according to the nutrition program of Burkina Faso.

Trial site selection The study will take place in Nanoro,Burkina Faso.

Recruitment and retention Prior to SMC first Round, children under five years living across HDSS area will be identified from the dataset of the last update round. Potential study participants will be randomly drawn from this list of children. Home visit will be performed to confirm the presence of the child, notify and inform parents of eligible participants about study and where possible obtain informed consent. Absent children or children whose parents are not willing to participate, will not be considered and will be replaced by other eligible children from the list. Children will be included after confirmation of the administration of the first dose of SMC Round 1 and after written consent is provided by the parents or guardians. Included children will be randomly allocated to one of the three study arms: (i) SMC + Vitamin A alone (ii) SMC+ Vitamin A+ Zinc and (iii) SMC+ Vitamin A + Plumpy'Doz. In case of many eligible children within a household, only one child will be included in order to avoid contamination between test and control groups. The randomized children will be followed-up actively for six Months and passively for six the next six months.

Trial subject safety All the products that will be used in this study are recommended by WHO and are already used as part of routine management of acute malnutrition in Burkina Faso.

Health service research issues, health economics and/or quality of life measures The project will promote economic development and welfare in Burkina Faso: the outcomes of this project will contribute indirectly to the economic development by reducing the burden of malaria and malnutrition, which constitute significant threats to economic development in the country.

Patient and/or community involvement The project will involve key stakeholders (Household and families of children, community health workers, health professionals, policy makers and representative of local community) at all levels of the health system in Burkina Faso through regular meetings.

Trial Steering Committee Prior to the study start, a trial steering committee will be set. This committee will comprise five independent members: a pediatrician, a nutritionist, a member of the Nanoro health district executive team, representatives of the national malaria and nutrition programs. The committee will monitor the progress of the trial through regular teleconferences and physical meetings (twice during the course of the intervention), advice on the scientific credibility and on specific issues that may arise during the course of the study. All decisions taken by this committee will be made by majority vote and will be documented.

Data Safety Management Board (DSMB) There will be no DSMB. Regular feedback on the effectiveness and safety of the combined intervention will be made available to local and national drug regulatory authorities within the Nanoro site and at the country level. When children under SMC coverage are missed, local health authorities will be informed immediately.

Trial Monitoring IRSS will contract an independent monitor and ensure that the study is adequately monitored. The monitor will verify the best conduct of the study through phone calls with the principal investigator and other study staff. Two monitoring visits are planned: an initiation visit before the enrolment of the first participant and a close-out visit after the last patient has completed the follow-up.

Ethical and regulatory approval The study protocol will have the approval of the Ethics Committees for Health Research in Burkina Faso prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Children under SMC coverage (6-59months old),
* living within the HDSS coverage area,
* ability to complete the study follow-up period,
* written consent obtained from parents

Exclusion Criteria:

* individual not under SMC coverage,
* Children under SMC coverage who did not receive the treatment (Amodiaquine-Sulfadoxine-Pyrimethamine) or the Vitamin Supplementation,
* ill individual at the time of the enrolment including uncomplicated/severe malaria or severe malnutrition,
* known allergy to Vitamin A or Zinc or Plumpy'Doz,
* planned travel or inability to complete the study follow-up,
* and unwillingness to participate to the study.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1059 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-07-04 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
The relative risk of the incidence of clinical malaria | One year
  The ration of the number of malaria cases in intervention over comparator arm hospitalisation and mortality in SMC group compared to SMC + supplement groups
The mid-upper arm circumference gain | One year
  The difference between baseline MUAC and MUAC at the end of the study period in the intervention groups compared to the control group
Weight gain | One year
  Difference between weight at baseline and weight at the end of the study
prevalence of anemia | one year
  prevalence of anemia in each arm

SECONDARY OUTCOMES:
The prevalence of mutant pfcrt allele | One year
  Difference between prevalence of mutant pfcrt in pre and post intervention months study period in malaria positive sample
The prevalence of mutant pfmdr1 allele | One year
  Difference between prevalence of mutant pfmdr1 in pre and post intervention months study period in malaria positive sample
The prevalence of mutant dhfr allele | One year
  Difference between prevalence of mutant dhfr in pre and post intervention months study period in malaria positive sample
The prevalence of mutant dhps allele | One year
  Difference between prevalence of mutant dhps in pre and post intervention months study period in malaria positive sample
SMC coverage | Six months
  SMC coverage in the area will be determined as the ratio of children who actually received the intervention to the predetermined sample of eligible children from the HDSS dataset.
SMC Compliance | Six months
  proportion of full compliant individual over the total per arm the predetermined sample of eligible children from the HDSS dataset. Compliance will be determined by calculating, for each participant, the ratio between the number of tablets / packets taken and the number of tablets / packets that the patient should have taken. Two groups of participants will be described: compliant = 100% treatment compliance and non-compliant = other cases
The incidence of adverse events in each study group will be considered | Six months
  The number of adverse events in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche en Sciences de la Santé/ Clinical Research Unit of Nanoro, Ouagadougou, Kadiogo, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Data on Plasmodium resistance will be shared with Infectious Diseases Data Observatory (IDDO)/ WorldWide Antimalarial Resistance Network (WWARN). The WHO will have access to the data to facilitate the development of new malaria control policy. Data will be made available to partners and as well as for other interested groups through the IDDO platform.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared within a year after database lock for unlimited time
Access Criteria: free access

REFERENCES:
- [Derived] Sondo P, Kabore B, Rouamba T, Compaore E, Tibiri YNG, Kabore HALF, Derra K, Tahita MC, Ilboudo H, Tougri G, Bouda I, Dakyo T, Kafando H, Ouedraogo F, Rouamba E, Hien SF, Kazienga A, Compaore CS, Bambara E, Nana M, Dahal P, Garanet F, Kabore W, Lefevre T, Guerin P, Tinto H. Enhanced effect of seasonal malaria chemoprevention when coupled with nutrients supplementation for preventing malaria in children under 5 years old in Burkina Faso: a randomized open label trial. Malar J. 2023 Oct 18;22(1):315. doi: 10.1186/s12936-023-04745-6. PMID 37853408
- [Derived] Sondo P, Tahita MC, Rouamba T, Derra K, Kabore B, Compaore CS, Ouedraogo F, Rouamba E, Ilboudo H, Bambara EA, Nana M, Sawadogo EY, Sorgho H, Some AM, Valea I, Dahal P, Traore/Coulibaly M, Tinto H. Assessment of a combined strategy of seasonal malaria chemoprevention and supplementation with vitamin A, zinc and Plumpy'Doz to prevent malaria and malnutrition in children under 5 years old in Burkina Faso: a randomized open-label trial (SMC-NUT). Trials. 2021 May 24;22(1):360. doi: 10.1186/s13063-021-05320-7. PMID 34030705